CLINICAL TRIAL: NCT04986098
Title: Clinical Study on the Effectiveness and Safety Evaluation of Directional Atherectomy Combined With Drug-coated Balloons in the Treatment of Femoral Popliteal Artery Occlusion
Brief Title: Clinical Study on the Effectiveness and Safety Evaluation of Directional Atherectomy Combined With Drug-coated Balloons
Acronym: Remove
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: Hongfei Sang
Record Dates: First submitted 2021-07-12; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

INTERVENTIONS:
Device: TurboHawk — Directly remove the diseased plaque in the blood vessel to increase the effective lumen in the blood vessel
Drug: Paclitaxel — Paclitaxel

SUMMARY:
DCB can maximize the patency rate of blood vessels on the basis of intraluminal DA. DA+DCB treatment is effective and safe [8], and the advantages of DA and DCB in the treatment of severe calcification and occlusive disease across joints and lower extremities have been confirmed. The combined application of DA and DCB in the treatment of peripheral arterial disease has a good early and mid-term effect. Konstantinos et al. reported that DARRT has a higher first-phase patency rate compared with DCB. A retrospective study by Sebastian et al. showed that compared with PTA after DA, the combination of DA and DCB has a better event-free survival rate after 12 months of follow-up. Therefore, DA combined with DCB therapy may be one of the best and most promising methods for the treatment of lower extremity ASO.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Ruthford grade 2-5 patients
* For patients whose arteries in both lower extremities meet the enrollment criteria, both lower extremities can be included
* At least one outflow tract over 10 cm at the distal end of the knee is continuous with a healthy back of the foot or internal and external arteries of the plantar
* The guide wire clearly passed through the lesion and the follow-up treatment was performed. In the case of failed anterograde passage, reverse puncture to achieve the guide wire through the lesion can also be included in the group
* After the failure of the first intracavitary treatment, the blood vessel can be recanalized by the intracavitary treatment again, and it can still be included in the group
* Patients with aortic iliac artery disease can be included in the group after the aortic artery is opened
* Patients who are willing to participate in this study and sign informed consent
* For severely infected R6 patients, if the infection is effectively controlled, they can be considered for inclusion

Exclusion Criteria:

* Patients who refuse to participate in this observational study
* Femoral popliteal artery disease with acute and subacute thrombosis
* Patients with thromboangiitis
* Patients who have failed endovascular treatment and transferred to surgical treatment
* For patients who have received plaque exfoliation on the femoral artery
* Patients who are allergic to heparin, low molecular weight heparin and contrast agents
* Patients enrolled in other clinical studies in the past 3 months
* Pregnant women
* Patients who have a life span of less than 2 years due to serious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASO patients with femoral popliteal artery occlusion
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary vascular patency rate | 24 months
  Free-Target lesion reconstruction rate（F-TLR）at 24 months after operation
Major adverse event | 24 months
  MAE within 24 months after surgery

SECONDARY OUTCOMES:
Quality of life assessment | 24 months
  Quality of life assessment (VAS-QOL) after discharge, 1, 3, 6, 12, and 24 months after operation
ABI | 24 months
  Ankle-brachial index (ABI) at discharge, 1, 3, 6, 12, and 24 months after operation
Rutherford classification | 24 months
  Discharge, 1, 3, 6, 12, and 24 months after the Rutherford classification
TLR | 24 months
  The incidence of TLR after discharge, 1, 3, 6, 12, and 24 months
TVR | 24 months
  The incidence of TVR after discharge, 1, 3, 6, 12, and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided